CLINICAL TRIAL: NCT04134364
Title: The Effect of 3-day Oral Administration of Lamina-G on Epigastric Pain or Soreness After Gastric Biopsy
Brief Title: The Effect of Lamina-G on Gastrointestinal Symptom After Gastric Biopsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Su Youn Nam, Assistant Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KNUMC 2016-02-002
Record Dates: First submitted 2019-09-14; First posted 2019-10-22 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Gastrointestinal Symptom
MeSH Terms: interventions — Alginates

STUDY DESIGN:
Intervention Model Description: open labeled, single-center randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): no medication after gastric biopsy
- treatment (Experimental): oral administration of sodium alginate (LaminaG) after gastric biopsy
  Interventions: Drug: Sodium alginate

INTERVENTIONS:
Drug: Sodium alginate — 3 days oral administration of sodium alginate after gastric biopsy
  Arms: treatment

SUMMARY:
Sometimes, subjects complain about gastrointestinal symptoms after esophagogastroduodenoscopy and biopsy. The aim of this study is to investigate the effect of sodium alginate (Lamina-G®) on biopsy-related gastrointestinal symptom.

DETAILED DESCRIPTION:
This study is an open labeled, single-center randomized controlled trials. Patients who underwent upper enoscopy with biopsy were randomly assigned to medication and control group. In the medication group, sodium alginate was administered after EGD during 3 days. All patients underwent a questionnaire to check the presence of gastrointestinal symptoms at baseline and on the day after return home. After 3 days, gastrointestinal symptoms were investigated by telephone survey. Gastrointestinal symptom was scaled by upper gastrointestinal symptom rate score (GSRS). Upper GSRS contains 8 items and 3 scales; abdominal pain (abdominal pain, epigastric pain/hunger soreness, nausea), reflux symptom (Heartburn/reflux/belching gas), indigestion symptom (abdominal distension, borborygmus).

ELIGIBILITY:
Inclusion Criteria:

Age from 18 to 80 years Persons who assigned on the written consent for the clinical trial. Persons who underwent upper endoscopy and gastric biopsy

Exclusion Criteria:

Gastrectomy Severe cardiovascular, pulmonary, or endocrine disease Renal or hepatic dysfunction Hematologic disease Gastric cancer Active peptic ulcer User of proton pump inhibitor, H2 blocker, mucoprotectant Immediate significant bleeding after biopsy Pregnant women Allergy history for sodium alginate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
gastrointestinal symptom | baseline endoscopy (T0)
  Upper Gastrointestinal Symptom Rating Scale (8 domain) : score : 0,1,2,3 in each domain (0: none, 3: severe)
gastrointestinal symptom | within 24 hours after endoscopy (T1)
  Upper Gastrointestinal Symptom Rating Scale (8 domain) : score : 0,1,2,3 in each domain (0: none, 3: severe)
gastrointestinal symptom | 3 days after endoscopy (T3)
  Upper Gastrointestinal Symptom Rating Scale (8 domain) : score : 0,1,2,3 in each domain (0: none, 3: severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No